CLINICAL TRIAL: NCT06029413
Title: Myo Vs. Myofascial Injection for Myofascial Trigger Points. Is There Really a Difference? A Randomized Controlled Trial
Brief Title: Myo vs. Myofascial Injection for Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Buğra İnce, Assoc. Professor, MD, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOY23
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Myofascial Pain; Myofascial Trigger Point Pain; Trigger Point Pain, Myofascial
Keywords: usg-guided trigger point injections; myofascial pain; myofascial trigger point; fascial hydrodilatation
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: This study is planned to compare the effects of USG guided intramuscular trigger point injection with the effects of USG guided intramuscular plus fascial trigger point injection. This is a single-center randomized trial with 2 parallel arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research arm (Experimental): After the myofascial trigger points are determined by ultrasonography (HI VISION Preirus; Hitachi Aloka Medical, Ltd., Tokyo, Japan), injections will be given to the myofascial layers from the deep to the superficial. First, the local anesthetic solution will be injected to create a separation in the intermuscle (epimysial) fascia. The injectable will then be infiltrated into the intermuscular hypoechoic nodule. Then, the deep fascia will be infiltrated layer by layer. Finally, the procedure will be completed by infiltrating the superficial fascia.
  Interventions: Procedure: myo + fascial injection
- Control arm (Active Comparator): Patients in the control group will be injected with the same amount of local anesthetic solution under ultrasound guidance to intramuscular hypoechoic nodules detected by ultrasonography (HI VISION Preirus; Hitachi Aloka Medical, Ltd., Tokyo, Japan).
  Interventions: Procedure: traditional trigger point injection

INTERVENTIONS:
Procedure: myo + fascial injection — 10 cc 0.5 % lidocain solution injection for intermuscular hypersensitive nodule as well as for fascial layers as described.
  Arms: Research arm
Procedure: traditional trigger point injection — 10 cc 0.5 % lidocain solution injection for intermuscular hypersensitive nodule as described.
  Arms: Control arm

SUMMARY:
In this study, the effectiveness of two different application methods that can be used in myofascial trigger point injection treatment will be compared.

DETAILED DESCRIPTION:
This study aims to compare the intramuscular trigger point injection, which is traditionally used in the treatment of myofascial trigger points with the method in which facial layers are also included in the application.

ELIGIBILITY:
Inclusion Criteria:

Pain in the upper back area

Detection of active trigger point in upper back muscles (trapezius, levator scapula, rhomboids, supraspinatus and infraspinatus)

Presence of at least two of the three criteria recommended for the diagnosis of trigger point:

1. Taut band
2. Hypersensitive point
3. Referred pain

Pain VAS score ≥ 4

Between the ages of 18-65 -

Exclusion Criteria:

Using analgesics or anti-inflammatory medicines.

Having received physical therapy for the same symptoms in the past 3 months

Serious psychiatric illness

Presence of malignancy or infection

Coagulation disorder

Pregnancy

History of operation in the relevant region

Presence of fibromyalgia syndrome

History of allergy to local anesthetics

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
VAS(Visual Analog Scale) | Baseline
  Pain intensity will be evaluated with the visual analog scale (VAS). VAS is a scale used to digitize subjective values such as behavior or characteristics that cannot be measured directly. Two end definitions of the parameter to be evaluated are written on both ends of a 10 cm line and the patient is asked to indicate where his/her condition is appropriate on this line by drawing a line (0. : no pain, 10: very severe pain)
VAS(Visual Analog Scale) | 30 minutes after intervention
  Pain intensity will be evaluated with the visual analog scale (VAS). VAS is a scale used to digitize subjective values such as behavior or characteristics that cannot be measured directly. Two end definitions of the parameter to be evaluated are written on both ends of a 10 cm line and the patient is asked to indicate where his/her condition is appropriate on this line by drawing a line (0. : no pain, 10: very severe pain)
VAS(Visual Analog Scale) | 72 hours after intervention
  Pain intensity will be evaluated with the visual analog scale (VAS). VAS is a scale used to digitize subjective values such as behavior or characteristics that cannot be measured directly. Two end definitions of the parameter to be evaluated are written on both ends of a 10 cm line and the patient is asked to indicate where his/her condition is appropriate on this line by drawing a line (0. : no pain, 10: very severe pain)
VAS(Visual Analog Scale) | 1 week after intervention
  Pain intensity will be evaluated with the visual analog scale (VAS). VAS is a scale used to digitize subjective values such as behavior or characteristics that cannot be measured directly. Two end definitions of the parameter to be evaluated are written on both ends of a 10 cm line and the patient is asked to indicate where his/her condition is appropriate on this line by drawing a line (0. : no pain, 10: very severe pain)

SECONDARY OUTCOMES:
Pressure Pain Threshold | Baseline
  The Baseline 1200-303 (Push-Pull Force Gauge®, Fabrication Enterprises, Inc.) algometer will be used to measure pressure pain threshold. The Baseline 1200-3031 cm2 is a dynamometer applied with a flat tip. The device is brought into contact with the skin at an angle of 90º and a force is applied to provide an increase of 1 kg per second. The first value at which the patient feels the sensation of pain is recorded. The average of 3 measurements taken at 30-second intervals is recorded as the patient's pressure pain threshold
Pressure Pain Threshold | 30 minutes after intervention
  The Baseline 1200-303 (Push-Pull Force Gauge®, Fabrication Enterprises, Inc.) algometer will be used to measure pressure pain threshold. The Baseline 1200-3031 cm2 is a dynamometer applied with a flat tip. The device is brought into contact with the skin at an angle of 90º and a force is applied to provide an increase of 1 kg per second. The first value at which the patient feels the sensation of pain is recorded. The average of 3 measurements taken at 30-second intervals is recorded as the patient's pressure pain threshold
Pressure Pain Threshold | 72 hours after intervention
  The Baseline 1200-303 (Push-Pull Force Gauge®, Fabrication Enterprises, Inc.) algometer will be used to measure pressure pain threshold. The Baseline 1200-3031 cm2 is a dynamometer applied with a flat tip. The device is brought into contact with the skin at an angle of 90º and a force is applied to provide an increase of 1 kg per second. The first value at which the patient feels the sensation of pain is recorded. The average of 3 measurements taken at 30-second intervals is recorded as the patient's pressure pain threshold
Pressure Pain Threshold | 1 week after intervention
  The Baseline 1200-303 (Push-Pull Force Gauge®, Fabrication Enterprises, Inc.) algometer will be used to measure pressure pain threshold. The Baseline 1200-3031 cm2 is a dynamometer applied with a flat tip. The device is brought into contact with the skin at an angle of 90º and a force is applied to provide an increase of 1 kg per second. The first value at which the patient feels the sensation of pain is recorded. The average of 3 measurements taken at 30-second intervals is recorded as the patient's pressure pain threshold
Functional Status | Baseline
  The change in the functional status of the patients will be evaluated with the neck disability index (NDI). NDI is a 10-question questionnaire most commonly used to evaluate nonspecific mechanical neck pain. A total score between 0 and 50 is obtained by scoring each question between 0 (no disability) and 5 (complete disability). The validity and reliability study of the Turkish version of the scale was shown.
Functional Status | 72 hours after intervention
  The change in the functional status of the patients will be evaluated with the neck disability index (NDI). NDI is a 10-question questionnaire most commonly used to evaluate nonspecific mechanical neck pain. A total score between 0 and 50 is obtained by scoring each question between 0 (no disability) and 5 (complete disability). The validity and reliability study of the Turkish version of the scale was shown.
Functional Status | 1 week after intervention
  The change in the functional status of the patients will be evaluated with the neck disability index (NDI). NDI is a 10-question questionnaire most commonly used to evaluate nonspecific mechanical neck pain. A total score between 0 and 50 is obtained by scoring each question between 0 (no disability) and 5 (complete disability). The validity and reliability study of the Turkish version of the scale was shown.

CONTACTS AND LOCATIONS:
Overall Officials: Buğra İnce, Study Director — Izmir Bozyaka Education and Research Hospital
Locations (1):
- Izmir Bozyaka Education and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricci V, Ricci C, Mezian K, Nanka O, Ozcakar L. Trapezius Muscle and the Cutaneous Branches of Spinal Nerves: Sonographic/Anatomic Discussion of Myofascial Pain and Superficial Injections. Pain Med. 2023 Mar 1;24(3):221-225. doi: 10.1093/pm/pnac125. No abstract available. PMID 35980166
- [Background] Ricci V, Ricci C, Gervasoni F, Cocco G, Andreoli A, Ozcakar L. From Histoanatomy to Sonography in Myofascial Pain Syndrome: A EURO-MUSCULUS/USPRM Approach. Am J Phys Med Rehabil. 2023 Jan 1;102(1):92-97. doi: 10.1097/PHM.0000000000001975. Epub 2022 Jan 21. PMID 35067549
- [Background] Pirri C, Pirri N, Guidolin D, Macchi V, De Caro R, Stecco C. Ultrasound Imaging of the Superficial Fascia in the Upper Limb: Arm and Forearm. Diagnostics (Basel). 2022 Aug 4;12(8):1884. doi: 10.3390/diagnostics12081884. PMID 36010234
- [Background] Nouged E, Dajani J, Ku B, Al-Eryani K, Padilla M, Enciso R. Local Anesthetic Injections for the Short-Term Treatment of Head and Neck Myofascial Pain Syndrome: A Systematic Review with Meta-Analysis. J Oral Facial Pain Headache. 2019 Spring;33(2):183-198. doi: 10.11607/ofph.2277. Epub 2019 Mar 20. PMID 30893405
- [Background] Stecco C, Macchi V, Porzionato A, Duparc F, De Caro R. The fascia: the forgotten structure. Ital J Anat Embryol. 2011;116(3):127-38. PMID 22852442